CLINICAL TRIAL: NCT01843738
Title: Radiation Use During Vemurafenib and Cobimetinib Treatment in Patients With BRAFV600 Mutated Stage IV or Unresectable Stage III Melanoma
Brief Title: Radiation Use During Vemurafenib Treatment
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Competing Trials
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI64498; NCT02042040 (obsolete NCT alias)
Record Dates: First submitted 2013-04-19; First posted 2013-05-01 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: BRAFV600 Mutation; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Radiotherapy; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental)
  Interventions: Radiation: Radiation therapy; Drug: Vemurafenib

INTERVENTIONS:
Radiation: Radiation therapy — Per standard of care
Drug: Vemurafenib — The starting dose of vemurafenib will be the patient's baseline tolerating dose, between 720 - and 960 mg PO bid.

SUMMARY:
Patients are being asked to take part because they have melanoma that has spread to other organs in their body (metastatic). As part of this study, patients will receive radiation therapy and an approved drug (Vemurafenib).

DETAILED DESCRIPTION:
Patients will be treated with vemurafenib plus radiation therapy (RT) based upon the administration schedule. The starting dose of vemurafenib will be the patient's baseline tolerating dose, between 720 - and 960 mg by mouth. Patients must be tolerating at a minimum 720mg for one cycle (28 days) prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosis of BRAFV600 mutated Stage IV or unresectable Stage III melanoma
* Actively receiving treatment with vemurafenib as single agent and tolerating at least 720 mg bid for one cycle (28 days).
* In the opinion of the investigator, patients who are progressing in an area where radiation may provide benefit from either:

  * Symptom control
  * Oligo-progression, defined as progression in up to 3 areas where focal treatment would provide benefit.
* Patients with brain metastases will be allowed provided they meet all of the following criteria:

  * Small, < 1cm metastases which are untreated are allowed so long as in the opinion of the investigator they do not require immediate treatment by radiation or surgery
  * Asymptomatic, treated brain metastases which are stable for 4 weeks prior to study entry are allowed
  * If patients are requiring steroids for their brain metastases, they must be on a stable dose for two weeks prior to study entry, and maintain that steroid dosing during the radiation treatments
* Adequate bone marrow function as defined by: ANC > 1.0 k/uL, Platelets > 75 k/uL, Hemoglobin > 8 g/dL
* Adequate hepatic function: Total bilirubin < 1.5 times the institutional upper limit of normal, ALT/AST < 2.5 times the institutional upper limit of normal
* Adequate renal function as defined by serum creatinin < 1.5 times the upper limit of normal.
* Negative serum pregnancy test at screening for women of child bearing potential within 10 days of starting vemurafenib treatment . Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for > 1 year
* Fertile men and women must agree to use an acceptable method of birth control during treatment and for at least 2 months after discontinuation of vemurafenib.
* Able and willing to provide informed consent to an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Screening QTc interval > 450 msec on EKG
* Known HIV positivity or AIDS-related illness, or active HBV, or active HCV.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, serious cardiac arrhythmia requiring medication, uncontrolled hypertension, cerebrovascular accident or transient ischemic attack, or symptomatic pulmonary embolism.
* Malabsorption disorder that would preclude adequate vemurafenib absorption.
* Other medical condition present that in the opinion of the investigator will hinder the subjects ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | 36 months
  To evaluate the safety of radiation combined with vemurafenib treatment in patients with BRAFV600 mutated Stage IV or unresectable Stage III melanoma

SECONDARY OUTCOMES:
Response rate | 36 months
  To evaluate response rates as assessed by RECIST criteria 1.1, at baseline, and at 8 week intervals throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Grossmann, MD, PhD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States